CLINICAL TRIAL: NCT00365898
Title: A Study of the Efficacy and Safety of 8 Mg Hydromorphone Hydrochloride Extended-Release Compared to Placebo in Subjects With Persistent Pain
Brief Title: Efficacy and Safety of Hydromorphone Hydrochloride Extended-Release Compared to Placebo in Subjects With Persistent Pain
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Purdue Pharma LP (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HMP3011
Record Dates: First submitted 2006-08-16; First posted 2006-08-18 (Estimated); Last update posted 2006-08-18 (Estimated); Status verified 2006-08

CONDITIONS: Chronic Non-Malignant Pain
Keywords: Chronic non-malignant pain, opioid

INTERVENTIONS:
Drug: Hydromorphone Hydrochloride Extended-Release

SUMMARY:
The objective of this study is to assess the efficacy and safety of 8 mg Hydromorphone Hydrochloride Extended-Release.

DETAILED DESCRIPTION:
The primary efficacy objective of this study is to compare the time to emergence of inadequate analgesia of 8 mg Hydromorphone Hydrochloride Extended-Release taken once every 24 hours versus placebo in the treatment of patients with persistent pain who require an opioid medication for control of their pain.

ELIGIBILITY:
Inclusion Criteria:

* persistent, moderate-to-severe noncancer related pain requiring continuous analgesia for weeks to months, or longer, who are currently taking 20 to 40 mg of oxycodone or opioid equivalents per day for control of their persistent pain and who are willing to accept the possibility of receiving placebo during the Double-Blind Phase

Exclusion Criteria:

* Patients already receiving opioid medication at an average total daily dose greater than 40 mg of oxycodone or opioid equivalents during the last week prior to study entry.

Other protocol-specific exclusion/inclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 380
Dates: Start 2005-07; Study Completion 2005-07

PRIMARY OUTCOMES:
Time to emergence of inadequate analgesia. Emergence of inadequate analgesia is defined as one or more of the following: a) the subject has a rating of poor or fair on the Patient Global Assessment of Pain Medicatio

SECONDARY OUTCOMES:
Patient Global Assessment of Pain Medication
Pain Control Questionnaire

CONTACTS AND LOCATIONS:
Locations (14):
- United States (14):
  - Arizona Research Center 2525 W. Greenway Rd. Suite 114, Phoenix, Arizona
  - Clinical Research of West Florida, Inc. 2147 NE Coachman Road, Clearwater, Florida
  - LCFP, Inc. 12631 World Plaza Lane Building 54, Fort Myers, Florida
  - Pharmaceutical Research Associates 1395 N. Courtenay Pkwy, Merritt Island, Florida
  - Stedman Clinical Trials 3212 Cove Bend Drive, Tampa, Florida
  - Palm Beach Research Center 1897 Palm Beach Lakes Blvd., West Palm Beach, Florida
  - Gold Coast Research 2965 Surrey Lane, Weston, Florida
  - PharmQuest 301 E Wendover Avenue Suite 411, Greensboro, North Carolina
  - Hightop Medical Research Center 6103 Hamilton Anenue, Cincinnati, Ohio
  - Research Institute of Greater Dayton 1010 Woodman Drive, Dayton, Ohio
  - Pharmacotherapy Research Associates, Inc. 3620 Court Drive, Zanesville, Ohio
  - Allegheny Pain Management-PC 1402 Ninth Ave, Altoona, Pennsylvania
  - he Tipton Medical & Diagnostic Center #334 Route 220, Tipton, Pennsylvania
  - Preferred Primary Care Physicians 202 Jacob Murphy Lane, Uniontown, Pennsylvania